CLINICAL TRIAL: NCT05263856
Title: The Effect of Laser Acupuncture Intervention to the Prognosis After Total Knee Replacement (TKR) Surgery
Brief Title: The Effect of Laser Acupuncture Intervention to the Prognosis After TKR Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH111-REC2-026; 1-CMUBHR109-005 (Other: China Medical University Beigang Hospital)
Record Dates: First submitted 2022-02-10; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Knee Osteoarthritis; Total Knee Replacement
Keywords: laser acupuncture; low level laser therapy; total knee replacement; myofascial trigger point; auricular acupuncture
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser acupuncture intervention (Experimental): In this arm, subjects will receive laser acupuncture (LA) intervention during hospitalization after total knee replacement (TKR) surgery until discharge once a day. LA will stimulate on the 1) bilateral reflection areas of ear associated knee and pain mechanism, including Knee, Sympathetic Autonomic, Zero, Thalamus, Master Cerebral, Master Sensorial points, with 6 points unilaterl and 12 points in total, and 2) myofascial trigger point around knee joint, which may affect function performance and prognosis after TKR, including quadriceps, tensor fascia lata,adductor major,sartorius, hamstrings, gastrocnemius muscles, with 10 points in total.
  Interventions: Device: laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — The parameter setting of 810nm wavelength laser acupuncture device in 1) ear were irradiated with a 4mm probe, adjusted to Nogier A frequency for acute treatment, and the pulsed mode was irradiated with an emission frequency of 200mW for 10seconds, each acupoint provided 1 joule of energy with total of 12joules,and 2) myofascial trigger point were irradiated with a 10mm probe, adjusted to Nogier C frequency for muscle treatment, and the pulsed mode was irradiated with an emission frequency of 500mW for 20 seconds, each acupoint provided 5 joule of energy with total of 50 joules, providing a total of 62 joules of one intervention session.
  Other Names: low level laser therapy

SUMMARY:
This study protocol is mainly focus on the patients, who suffer pain, swelling, or range of motion limitation after total knee replacement (TKR) surgery procedure,would be relieved by use non-invasive laser acupuncture to stimuli on 1) the reflection areas of ear acupuncture point associated knee and pain mechanism; 2) muscle trigger points around knee joint with adequate frequency and energy power to stimuli.

DETAILED DESCRIPTION:
Traditional Chinese acupuncture has a history of several thousand years. The World Health Organization has published guidelines describing the efficacy of acupuncture in the cure or relief of 64 different symptoms and conditions as one of the most representative intangible cultural heritage of humanity. However, for the need of patients and the gradual progress of technology, the applications of laser acupuncture become widespread. Laser acupuncture (LA) is not only applicated to stimuli specific areas in need, but also one of non-invasive intervention technic with hurtless intervention, no hematoma, bleeding or swelling unpleasant feeling after intervention, which could be more accepted by children, weakness people, and patients who afraid of acupuncture. To the area that traditional Chinese acupuncture could not stimuli easily of some area reflect to brain precisely, laser acupuncture is comparably convenient to supply adaptive energy input.

The goals of this study protocol is focus on the patients who accept total knee replacement (TKR), who usually suffer pain, swelling, or range of motion limitation after TKR surgery procedure, and the investigators want to use non-invasive LA to stimuli on 1) the reflection areas of ear acupuncture point associated knee and pain mechanism; 2) myofascial trigger points around knee joint, which may affect functional performance and prognosis after TKR procedure, with adequate frequency and energy power to stimuli, to observe the efficacy of LA on pain relief, swelling decline, and range of motion in knee joint improvement. One the one side, the investigators want to shorten the period of recovery, accelerate the function performance, and enhance the quality of life of patients after TKR procedure by LA intervention,on the other side, the investigators also want to confirm the value and curative effect of LA on clinical application and to evoke new idea for further development to traditional Chinese acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients who completed total knee replacement (TKR) during hospitalization
* Understands and obeys conventional treatment instructions
* Subjects who are willing to receive laser acupuncture treatment

Exclusion Criteria:

* There are contraindications to general treatment, such as serious medical problems, recent serious trauma, or pregnant and lactated women.
* There has been a history of drug abuse (including excess alcohol) that affects pain assessment.
* Infection, ulcer or injury on the local skin surface at the intervention site
* Aphasia, inability to answer questions
* Cognitive impairment, unable to cooperate with the experiment

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes from Visual Analog Scale for myofascial trigger points | The 1 day Before the first laser acupuncture and the 1 day after the last laser acupuncture intervention
  A Visual Analog Scale consists of a line, often 10 cm long, with verbal anchors at either end, on left of line, zero, meant no pain otherwise on right, 10, meant strong pain. The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.
Changes from WOMAC scale of Knee (modified in Chinese) | Baseline (Before surgery), 1 month after surgery, and 3 months after surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Knee and other osteoarthritis. This modified version is a self-administered questionnaire consisting into 4 subscales and mainly focus on functional performance: pain and ability to walk, pain and ability to go up and down stairs, knee swelling, and the range of motion of knee flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chuan Chang, M.D., Principal Investigator — China Medical University Beigang Hospital
Locations (1):
- China Medical University Beigang Hospital, Beigang, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided